CLINICAL TRIAL: NCT01931124
Title: Effect of High Intensity and Moderate Training on Maximal Oxygen Uptake and Activity Levels in an Elderly Norwegian Population
Brief Title: High Intensity and Moderate Training and Maximal Oxygen Uptake and Activity Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gen100sub4
Record Dates: First submitted 2013-07-19; First posted 2013-08-29 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Ageing
Keywords: maximal oxygen uptake, activity levels, elderly
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Training (Experimental): training at high intensities ranging from 85-95% of maximal heart rate
  Interventions: Behavioral: High Intensity Training
- Moderate Intensity Training (Experimental): training at intensities of 65-75% of maximal heart rate
  Interventions: Behavioral: Moderate Intensity Training

INTERVENTIONS:
Behavioral: High Intensity Training
  Arms: High Intensity Training
Behavioral: Moderate Intensity Training
  Arms: Moderate Intensity Training

SUMMARY:
Aim of the study is to investigate the effect of different types of training (high intensity and moderate training) on maximal oxygen uptake and activity levels in an elderly Norwegian population after one year training intervention. Baseline data include the activity levels assessed through self reported means as well as objectively measured activity data using activity monitors.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk at least 1km,
* born in 1938,1939,1940,1941 or 1942
* Sufficiently good health to be able to take part in the study, as determined by the researchers

Exclusion Criteria:

* Illness or disability that precludes exercise or hinders completion of the study
* Uncontrolled hypertension
* Symptomatic valve disease, hyper tropic cardio-myopathy or unstable angina
* Active cancer
* Test results indicating that study participation is unsafe
* Inclusion in other studies conflicting with participation in this one

Ages: 70 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1576 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
maximal oxygen uptake | 1 year
activity level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: dorthe stensvold, PhD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway